CLINICAL TRIAL: NCT06754215
Title: Development of a Contextually Tailored and Optimized Smoking Cessation Intervention for Homeless Youth
Brief Title: Smoking Cessation Intervention Development for Homeless Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: OSU-17281; NCI-2019-02248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K07CA216321 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Focus Groups; Interviews as Topic; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MOST STEP Ia (interview) (Experimental): Participants attend a semi-structured interview over 60 minutes to help establish theoretical model of contextually tailored smoking cessation for homeless youth.
  Interventions: Other: Interview
- MOST STEP Ib (survey) (Experimental): Participants complete a survey to help establish theoretical model of contextually tailored smoking cessation for homeless youth.
  Interventions: Other: Survey Administration
- MOST STEP II (feasibility study) (Experimental): Intervention components are identified and selected from Focus Groups. Participants take part in a study to assess these components for feasibility in implementing in coordination with homeless youth services, as well as determining main effect estimates for future studies.
  Interventions: Behavioral: Smoking Cessation Intervention
- MOST STEP II (focus groups) (Experimental): Participants attend focus groups to help identify a set of cessation intervention components for homeless youth and determine component acceptability and feasibility.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Participate in focus group
  Arms: MOST STEP II (focus groups)
Other: Interview — Participate in semi-structured interview
  Arms: MOST STEP Ia (interview)
Behavioral: Smoking Cessation Intervention — Participate in feasibility study of intervention components
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: MOST STEP II (feasibility study)
Other: Survey Administration — Complete survey
  Arms: MOST STEP Ib (survey)

SUMMARY:
This trial develops a contextually tailored and optimized smoking cessation intervention and studies smoking motivations and motivations to quit smoking in homeless youth. Identifying motivations for smoking and motivations to quit smoking may help researchers build a program to help homeless young people quit smoking cigarettes if desired.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish a theoretical framework for cessation among homeless youth incorporating phase-specific capabilities and opportunities impacting motivation to engage in cessation. (Multiphase Optimization STrategy [MOST] Step 1) II. Guided by the theoretical framework for cessation among homeless youth, identify a set of cessation intervention components and assess their implementation feasibility. (MOST Step 2)

OUTLINE:

MOST STEP Ia: Participants attend a semi-structured interview over 60 minutes to help establish theoretical model of contextually tailored smoking cessation for homeless youth.

MOST STEP Ib: Participants complete a survey to help establish theoretical model of contextually tailored smoking cessation for homeless youth.

MOST STEP II (FOCUS GROUPS): Participants attend focus groups to help identify a set of cessation intervention components for homeless youth and determine component acceptability and feasibility.

MOST STEP II (FEASIBILITY STUDY): Intervention components are identified and selected from Focus Groups. Participants take part in a study to assess these components for feasibility in implementing in coordination with homeless youth services, as well as determining main effect estimates for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Youth who report having smoked some or every day in the past week.
* Youth who meet criteria for homelessness defined by the 2002 McKinney-Vento Act including those who lack a fixed, regular, and adequate nighttime residence; live in a welfare hotel, or place without regular sleeping accommodations; or live in a shared residence with other persons due to the loss of one's housing or economic hardship.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 298 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Youth's psychological and physical capacity (capability) | Up to 3 years
  Participant's psychological and physical capacity that have prompted them in the past or may motivate them to 1) smoke, 2) make a quit attempt, and 3) engage in supported cessation will be captured. An iterative approach to team-based codebook development and coding will be used to analyze interview data. In Stage 1, text will be coded according to the specific research question using structural codes. In Stage 2, in depth codes will be created using emergent themes from the structurally coded text. The coders will create as many in depth codes as needed in order to capture all aspects of youth's perspective on current psychosocial influences on smoking, and the psychological and physical capacities critical to engagement in tobacco cessation intervention. Data is separated by the age cut-off for standard recommendations regarding cessation intervention (14-17 and 18-24) to assess if differences exist that should be considered for intervention in homeless drop in centers.
Youth's physical and social factors (opportunity) | Up to 3 years
  Participant's physical and social factors (opportunity) that have prompted them in the past or may motivate them to 1) smoke, 2) make a quit attempt, and 3) engage in supported cessation will be captured. In Stage 1, text will be coded according to the specific research question using structural codes. In Stage 2, in depth codes will be created using emergent themes from the structurally coded text. The coders will create as many in depth codes as needed in order to capture all aspects of youth's perspective on current psychosocial influences on smoking, and the physical and social opportunities critical to engagement in tobacco cessation intervention. Data is separated by the age cut-off for standard recommendations regarding cessation intervention (14-17 and 18-24) to assess if differences exist that should be considered for intervention in homeless drop in centers.

CONTACTS AND LOCATIONS:
Overall Officials: Julianna Nemeth, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu